CLINICAL TRIAL: NCT02816892
Title: Significance of Serum Tenascin C in Patients With Acute Aortic Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, CHAI Xiangping, Vice Director of emergency department，director of hospital office, Central South University
Other Study IDs: 2XY-ED-002
Record Dates: First submitted 2016-04-25; First posted 2016-06-29 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Aortic Dissection
Keywords: aortic dissection; biomarkers; diagnosis
MeSH Terms: conditions — Aortic Dissection; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Rupture group: Rupture was defined by direct visualisation of the discontinuity of the aortic wall by computed tomography, sonography, intraoperative findings or at autopsy with detection of blood in the pleural, pericardial or abdominal cavity.
- Covert rupture group: Covert rupture was defined as an intramural haematoma without detection of free blood in the body cavities.
- Acute dissection group: Acute dissection was defined when blood separating the layers of the aortic media was newly diagnosed.
- Chronic dissection group: Chronic dissection was defined as the absence of any visible propagation of a known dissection compared to preexisting examinations.
- Ectatic aneurysm group: Ectatic aneurysm was defined as a permanent localised dilatation of the aorta with a diameter of at least 50% greater than normal

SUMMARY:
This study aims to investigate Serum Tenascin C levels in patients with acute symptoms relating to a known or newly diagnosed aortic aneurysm in emergency department and reveals the possible role of Tenascin C in the development of the disease.

DETAILED DESCRIPTION:
Patients with acute and chronic aortic disease /survivors and non-survivors were compared. Further subgroup analysis on the characteristics of the aneurysm and patients were performed. The aneurysms (ruptured and dissected) were divided according to the style of the Stanford classification,according to the location of the pathology in aneurysms of the ascending thoracic aorta .the descending thoracic aorta, or the abdominal aorta.The subgroup were divided according to the extent of propagation of the disease (rupture,covered rupture, acute dissection, chronic dissection and ectasia). Rupture was defined by direct visualisation of the discontinuity of the aortic wall by computed tomography, sonography, intraoperative findings or at autopsy with detection of blood in the pleural, pericardial or abdominal cavity. Covert rupture was defined as an intramural haematoma without detection of free blood in the body cavities. Acute dissection was defined when blood separating the layers of the aortic media was newly diagnosed. Chronic dissection was defined as the absence of any visible propagation of a known dissection compared to preexisting examinations. Ectatic aneurysm was defined as a permanent localised dilatation of the aorta with a diameter of at least 50% greater than normal. Documentation of the surgical interventions and autopsy reports was used to confirm the diagnosis. In all patients the investigators collected the history, age of the patients, duration of pain, blood pressure at admission and laboratory parameters (haematocrit, creatinine) and Tenascin C Serum levels after admission to our emergency department immediately. The patients were followed up until hospital discharge and the outcome (survived/died) was recorded.

ELIGIBILITY:
Inclusion Criteria:

* adults
* sudden severe thoracic or abdominal pain

Exclusion Criteria:

* lesser than 18 years
* pregnant women
* trauma
* tumour

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who were suspected acute aortic disease in emergency department of the second xiangya hospital.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The level of serum tenascin-C | lesser than 48hours
  serum tenascin-C in ng/ml was measured by elasia

SECONDARY OUTCOMES:
Characteristics of enrolled subjects | lesser than 48hours
  age in years,sex,IBM in kg/m^2 and associated history was collected
The level of D-D，C-reactive protein，elastic protein fragment | lesser than 48hours
  The level of D-D in ng/ml，C-reactive proteinin ng/ml，elastic protein fragmentin ng/ml was measured by elasia

CONTACTS AND LOCATIONS:
Overall Officials: Xiangping Chai, M.D., Study Chair — Second Xiangya Hospital of Central South University
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes